CLINICAL TRIAL: NCT05580289
Title: The Effect of Local Dry Heat Applıcatıon and Half Shower on The Development of Postoperative Urinary Retentıon and Paın ın Patıents Applıed With Spınal Anesthesıa
Brief Title: The Effect of Local Dry Heat Applıcatıon and Half Shower on The Development of Urinary Retentıon and Paın
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Duzce-atiye-02
Record Dates: First submitted 2022-09-15; First posted 2022-10-14 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Spinal Anesthesia; Nursing; Bladder Retention; Dry Heat Application; Half Shower; Pain
MeSH Terms: conditions — Urinary Retention; Pain

STUDY DESIGN:
Intervention Model Description: randomised
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Routine care of the patient will be done and the level of pain will be determined with McGill pain scale questionnaire short form
- detrimental group (Experimental): Warm half shower + dry hot application will be applied to the experimental group in the early postoperative period.mplementation Phase: After mobilizing the patients in the experimental group, who have regained their muscle strength and can be mobilized, their legs will be washed with 40-45oC warm tap water for 5 minutes (down from the hip level) until their legs are up to the femur acetabulum level, and then the patient will be taken to the bed for 20 minutes. Dry hot application will be done over the bladder. Palpation and bladder examination will be performed every hour to understand bladder filling in patients who will be expected to urinate within 6-8 hours after surgery.
  Interventions: Other: half-shower and hot pack

INTERVENTIONS:
Other: half-shower and hot pack — The patients in the experimental group will be given hot application and half shower applications and the pain levels of the patients and the development of bladder retention will be followed.
  Arms: detrimental group

SUMMARY:
Urinary retention is defined as the inability to empty the bladder spontaneously even though the bladder is full. Although urinary retention is seen in two forms as acute and chronic, acute urinary retention is defined by the International Continence Society (ICS) as the situation where the patient is unable to urinate, the bladder is felt when palpated by hand, and the bladder content contains at least 150 ml of urine with pain. Chronic bladder retention is defined by ICS as a painless condition that can be felt when the bladder is palpated manually after urinating, with at least 150 ml of urine in the bladder content.

aim:The aim of this study is to determine the Effect of Postoperative Local Dry Hot Application and Half Shower Application on the Development of Bladder Retention and Pain in Patients undergoing Spinal Anesthesia.

DETAILED DESCRIPTION:
Urinary retention is defined as the inability to empty the bladder spontaneously even though the bladder is full. Although urinary retention is seen in two forms as acute and chronic, acute urinary retention is defined by the International Continence Society (ICS) as the situation where the patient is unable to urinate, the bladder is felt when palpated by hand, and the bladder content contains at least 150 ml of urine with pain. Chronic bladder retention is defined by ICS as a painless condition that can be felt when the bladder is palpated manually after urinating, with at least 150 ml of urine in the bladder content.

aim:The aim of this study is to determine the Effect of Postoperative Local Dry Hot Application and Half Shower Application on the Development of Bladder Retention and Pain in Patients undergoing Spinal Anesthesia.

methot : The study was planned as a single-blind randomized controlled experimental study with a parallel group design. In the study, half shower and dry hot application will be applied to the patients in the experimental group. On the other hand, the control group patients will not receive any intervention other than general treatment and care. Dry hot application and half shower application method used in the study is a method used routinely in nursing care. In this study, the effectiveness of this method, which is used routinely, will be tried to be demonstrated. Randomization will be done by block randomization method. Patients meeting the inclusion criteria will be assigned to the groups after obtaining their informed consent to accept the study. Assignment to groups will be made at randomizer.org.

In the analysis made in the G* power 3.1.9.7 program, it was determined that a total of 60 people should be reached. After the calculated sample size, 20% more of the sample will be included in the study in order to avoid the attrition bias. Therefore, it is aimed to complete the study with 72 patients.

There will be two groups as control and experimental groups in the research. Warm half shower + dry hot application will be applied to the experimental group in the early postoperative period, and the other group will be the control group, whose routine care will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Receiving spinal anesthesia
* Be over 18 years old
* Mobilize
* Agreeing to participate in the study voluntarily.
* To speak Turkish and to be able to read and write

Exclusion Criteria:

* Having any kidney disease
* Having a urological problem involving the bladder and urethra
* Not being able to mobilize
* Not being willing to participate in the study
* Presence of incision in the suprapubic region

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
bladder retention | one day
  The risk of developing bladder retention after surgery is expected to decrease in the experimental group compared to the post-intervention control group.
  We will use an implementation checking form that researchers prepare. İt contains every step related to research intervention such as bladder examination times, pain levels, etc.
  1. It will be decided that the patient can be mobilized after the surgery, and this process takes approximately 1 hour.
  2. It will be checked whether bladder retention has developed before the application.
  3. Hot application (20 minutes) and half shower (5 minutes) will be applied for a total of 25 minutes.
  4. It will be checked whether bladder retention develops after the application.
  5. Bladder palpation will be performed every hour until patients pass their first urination.
  This process will take approximately 6-8 hours.
pain level | one day
  Pain is expected to decrease in the experimental group compared to the control group after half-shower and hot application.
  Pain measurement will be made by McGill Pain Survey Short Form. The survey includes a visual analog score. The intensity of pain will measure the area in which the individual mark between 0 (no pain) and 10 (worst pain I felt in my life).
  The risk of developing pain after surgery is expected to change in the experimental group compared to the post-intervention control group.
  1. It will be decided that the patient can be mobilized after the surgery, and this process takes approximately 1 hour.
  2. It will be checked whether the pain has developed before the application.
  3. Hot application (20 minutes) and half shower (5 minutes) will be applied for a total of 25 minutes.
  4. It will be checked whether pain develops or pain level change after the application.
  5. Pain level will be performed every hour until patients pass their first urination.

CONTACTS AND LOCATIONS:
Overall Officials: esra yatkın, Principal Investigator — Duzce University
Locations (1):
- Duzce Univercity Medical Fauculty, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No